CLINICAL TRIAL: NCT04776421
Title: A Prospective Registration Study on Diverting Ileostomy and Anal Functional Outcomes After Anus Preservation Surgery in Middle and Low Rectal Cancer
Brief Title: Diverting Ileostomy and Anal Functional Outcomes After Anus Preservation Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Head of Department, The First Hospital of Jilin University
Other Study IDs: STARS-RC02
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Diverting Ileostomy; Middle and Low Rectal Cancer; Functional Outcome; Stoma Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ileostomy group
  Interventions: Procedure: Diverting ileostomy

INTERVENTIONS:
Procedure: Diverting ileostomy — Diverting ileostomy

SUMMARY:
Analyze the occurrence of complications, rectal function and quality of life after anus-preserving surgery for middle and low rectal cancer, so as to evaluate the role of protective ileostomy.

ELIGIBILITY:
Inclusion Criteria:

Necessary conditions: meet one of the following conditions

1. Difficult pelvis: narrow pelvis (diameter of ischial tuberosity <10 cm, diameter of ischial spine <12 cm) 13 or BMI≥30kg/m2 or tumor diameter≥5cm2.
2. To receive treatment before surgery: preoperative neoadjuvant radiotherapy or concurrent chemoradiation or ESD
3. The anastomosis is below the level of the levator ani muscle: such as ISR, TaTME surgery, etc.

Other conditions:

1. Age: 18 to 75 years old, male or female;
2. Preoperative biopsy pathological diagnosis of rectal adenocarcinoma;
3. Received MRI evaluation before surgery, and the distance between the lower edge of the tumor and the anal edge is no more than 10cm;
4. The clinical stage is T1-3N0-2M0;
5. Undertake elective laparoscopic TME for colon-rectal or colon-anal anastomosis
6. ECOG score 0-2;
7. Heart, lung, liver, and kidney functions can tolerate surgery;
8. Patients and their families can understand and are willing to participate in this clinical study, and sign informed consent.

Exclusion Criteria:

1. Past history of malignant colorectal tumors or recent diagnosis combined with other malignant tumors;
2. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. who need emergency surgery;
3. Neighboring organs need to be combined with organ removal
4. ASA grade ≥ grade IV and/or ECOG physical status score> 2 points;
5. Those who have severe liver and kidney function, cardiopulmonary function, blood coagulation dysfunction, or combined with serious underlying diseases that cannot tolerate surgery;
6. Have a history of severe mental illness;
7. Pregnant or lactating women;
8. Those with a history of taking hormone drugs;
9. Patients with other clinical and laboratory conditions considered by the investigator should not participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Middle and low rectal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
comprehensive complication index | 1 year
  comprehensive complication index, CCI

SECONDARY OUTCOMES:
Postoperative complications | 1 year
  Postoperative complications based on Clavien-Dindo
Incidence of anastomotic leakage | 1 year
Incidence of anastomotic stenosis | 1 year
Stoma-related complications | 3 months
Complications related to ileostomy reversal | three months after ileostomy reversal
Overall Survival | three years after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, Prof., Principal Investigator — Jilin University First Hospital

IPD SHARING:
Plan to Share IPD: No